CLINICAL TRIAL: NCT01657318
Title: A Prospective Observational Study on the Use of a Olivamine-containing Products in the Management of Patients With Compromised Nonhealing Lower Extremity Ulcers
Brief Title: Olivamine-containing Products in the Management of Patients With Nonhealing Lower Extremity Ulcers
Status: Terminated | Type: Observational
Why Stopped: challenges encountered in the methodology and concerns with the gold standard of treatment
Sponsor: De La Salle University Medical Center (Other)
Collaborators: Pinnaclife Inc. (Industry)
Responsible Party: Principal Investigator, Michael M. Lawenko MD, FPCS, Assistant Professor, De La Salle University Medical Center
Other Study IDs: AKMRC-12-004
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Ulcer; Skin Ulcer; Leg Ulcer; Diabetic Foot
Keywords: diabetic foot; leg ulcer
MeSH Terms: conditions — Ulcer; Skin Ulcer; Leg Ulcer; Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Wound Group: Treatment with Olivamine containing wound care products
  Interventions: Other: Olivamine containing wound care products

INTERVENTIONS:
Other: Olivamine containing wound care products — Continuous wound care with Olivamine containing products until wound closure. Intake of dietary supplement of 1 capsule for 60 days.
  Other Names: Olivamine Antiseptic Cleanser; Olivamine Cleansing Lotion; Olivamine Skin Restore Cream; Olivamine Wound Hydrogel; Miracle Olivamine Essential Dietary Supplement

SUMMARY:
In this study, the investigators hypothesize that the use of olivamine-containing products in the management of patients with compromised nonhealing lower extremity ulcers is feasible in the Philippine setting. It will result in complete ulcer healing or wound closure after 16 weeks.

DETAILED DESCRIPTION:
The specific aim of this study is to assess the feasibility of using olivamine-containing products in the management of patients with compromised nonhealing lower extremity ulcers in the Philippines. The primary endpoint of which is to evaluate the efficacy of Olivamine on healing of chronic lower extremity ulcers which will be assessed by rate of change in ulcer size (wound healing trajectory) and proportion with complete ulcer healing (wound closure) at 4, 8, 16 and 16 weeks compared to baseline, week 0.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years old or older.
* Patient has a diagnosis of arterial, diabetic foot, venous insufficiency, or pressure ulcer or surgical and traumatic wound.
* Patient's target study ulcer/wound is a lower extremity full thickness ulcer/wound not involving tendon, capsule, or bone.
* Patient's target study ulcer/wound and is ≥1.0 cm2 and ≤ 10.0 cm2 in size at the day of initial consult.
* Study ulcer/wound has been present for greater than 6 weeks prior to initial consult.
* Patients with Charcot foot deformities can be entered so long as the Charcot disease is not active, and the ulcer can be offloaded by an orthotic device.
* The patient has adequate circulation to the lower extremity as evidenced by an ABI (measured by Doppler) of ≥ 0.7. If the patient has non-compressible leg arteries, as documented by an ABI >1.3, then the patient must have a Toe-Brachial Index be > 0.6, or a toe pressure >50 mm Hg.
* Patient must have adequate in-home support to comply with all protocol-mandated visits and procedures, offloading or pressure redistribution as required, and proper application of study products and wound care regimen.
* Patient or his/her legal representative has read and signed the Institutional Review Board-approved Informed Consent form before Screening.

Exclusion Criteria:

* An ulcer/wound that is ≥10.0 cm2 and ≤ 1.0 cm2 in size at the day of initial consult is not eligible for this study.
* Patient has clinical evidence of gangrene or infection on any part of the affected foot.
* The patient is judged by the investigator or study staff to be unable or unlikely to comply with daily wound care instructions, or study visits.
* Patient has clinical evidence of active sepsis or invasive infection (e.g., cellulitis, osteomyelitis).
* Patient has muscle, tendon, or bone exposure in any ulcer bed.
* Patient has known sensitivity or allergy to any component of the study product - Olivamine10.
* Patient has one or more medical condition(s), including renal, hepatic, hematologic, neurologic, or immune disease that in the opinion of the - Investigator would make the patient an inappropriate candidate for this wound healing study.
* Patient has a malignant disease (other than squamous or basal cell carcinoma of the skin) not in remission for five years or more.
* Patient has known alcohol or drug abuse.
* Patient has a hematocrit greater than 60% or less than 27%.
* Patient's diabetes is under poor control as manifested by HbA1c of >10.0%.
* Patient has clinically significant renal insufficiency or creatinine greater than 2.0 mg/dL.
* Patient has chronic liver disease or clinically significant liver enzyme abnormality as evidenced by elevated AST, ALT, or bilirubin greater than 1.5 times upper limit of normal (ULN).
* Patient is receiving oral or parenteral corticosteroids, immunosuppressive or cytotoxic agents, or is anticipated to require such agents during the course of the study.
* Patient is using tobacco, or is exposed to a current smoker in their household. Patients may participate in the study if they have not used tobacco for 3 months and have not had a smoker in their household for 3 months.
* Patient is using any form of nicotine including nicotine patches, gums, or sprays.
* Patient has Acquired Immunodeficiency Syndrome (AIDS) or is known to be infected with Human Immunodeficiency Virus (HIV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential study subjects will be patients who are 18 years or older, has confirmed with the informed consent. He/she has a non-healing lower extremity ulcers compromised due to underlying factors such as peripheral arterial disease, diabetes, venous insufficiency, and pressure. The ulcer must be between 1.0 cm2 and 10 cm2.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2013-01-30 (Actual); Study Completion 2013-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Lawenko, MD, FPCS, Principal Investigator — De La Salle University Medical Center; Melchor V. Frias, MD, Study Chair — De La Salle Health Sciences Institute; Renato CA Ocampe, MD, FPCS, Study Director — De La Salle University Medical Center
Locations (1):
- De La Salle University Medical Center, Dasmariñas, Cavite, Philippines